CLINICAL TRIAL: NCT00121628
Title: A Phase 2, Open-label Study of AMG 706 to Treat Subjects With Locally Advanced or Metastatic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040273; NCT00331383 (obsolete NCT alias)
Record Dates: First submitted 2005-07-12; First posted 2005-07-21 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid cancer; Advanced thyroid cancer; Metastatic thyroid cancer; Medullary thyroid cancer; Follicular thyroid cancer; Papillary thyroid cancer; Hurthle cell thyroid cancer; Thyroid cancer treatments; Differentiated thyroid cancer and medullary thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Medullary; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid cancer, Hurthle cell | interventions — motesanib diphosphate

INTERVENTIONS:
Drug: AMG 706

SUMMARY:
The purpose of the study is to determine if AMG 706 will have clinically meaningful anti-tumor activity in subjects with locally advanced or metastatic thyroid cancer who are not candidates for radioactive iodine therapy or local therapies.

ELIGIBILITY:
Inclusion Criteria: - Histologically confirmed locally advanced or metastatic thyroid cancer - Measurable disease - Normal blood pressure (if history of hypertension, blood pressure must be controlled with medication) - Evidence of disease progression within 6 months before starting study (for differentiated thyroid cancer subjects) - Evidence of disease progression within 6 months before starting study OR symptomatic disease (for medullary thyroid cancer subjects) - Not a candidate for surgical resection, external beam radiotherapy, radioiodine therapy, or other local therapy - At least 18 years of age Exclusion Criteria: - Undifferentiated/anaplastic thyroid cancer - Untreated or symptomatic brain metastases - Prior malignancy, unless cured with treatment and no evidence of disease for greater than or equal to 3 years before starting study (history of thyroid cancer, in situ cervical cancer, or basal cell cancer of skin are exceptions) - Myocardial infarction or any unstable cardiac condition (e.g., congestive heart failure, unstable angina) within 1 year before starting study - Arterial thrombosis or deep vein thrombosis within 1 year before starting study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (complete response and partial response) as defined by modified RECIST

SECONDARY OUTCOMES:
Duration of response
Progression Free Survival
Changes in tumor markers
overall survival time
time to response
Tumour Related Symptoms (medullary thyroid cancer arm)
AMG 706 pharmacokinetic profile
patient reported outcome (EQ-5D)
Safety Endpoint: Incidence of treatment-emergent adverse events (including all, serious, treatment-related, and each by maximum severity).
Pharmacokinetic Enpoint: AMG 706 pharmacokinetic parameters (Cmax, t1/2, AUC0-24,C24)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Sherman SI, Wirth L, Droz J-P, Hofmann M, Bastholt L, Martins R, Licitra L, Eschenberg M, Sun Y-N, J
- [Derived] Bass MB, Sherman SI, Schlumberger MJ, Davis MT, Kivman L, Khoo HM, Notari KH, Peach M, Hei YJ, Patterson SD. Biomarkers as predictors of response to treatment with motesanib in patients with progressive advanced thyroid cancer. J Clin Endocrinol Metab. 2010 Nov;95(11):5018-27. doi: 10.1210/jc.2010-0947. Epub 2010 Aug 25. PMID 20739388
- [Derived] Sherman SI, Wirth LJ, Droz JP, Hofmann M, Bastholt L, Martins RG, Licitra L, Eschenberg MJ, Sun YN, Juan T, Stepan DE, Schlumberger MJ; Motesanib Thyroid Cancer Study Group. Motesanib diphosphate in progressive differentiated thyroid cancer. N Engl J Med. 2008 Jul 3;359(1):31-42. doi: 10.1056/NEJMoa075853. PMID 18596272
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com